CLINICAL TRIAL: NCT05566990
Title: A Multicenter, Open-Label, Phase III Study to Evaluate the Efficacy and Safety of LIV-GAMMA SN Inj.10% in Primary Immune Thrombocytopenia (ITP)
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of LIV-GAMMA SN Inj.10% in Primary Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Plasma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIg10%_ITP_III_2019
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIV-GAMMA SN Inj.10% (Experimental)
  Interventions: Biological: LIV-GAMMA SN Inj.10%

INTERVENTIONS:
Biological: LIV-GAMMA SN Inj.10% — LIV-GAMMA SN Inj. 10% is administered intravenously at a dose of 1 g/kg daily for 2 consecutive days to patients with primary immune thrombocytopenia.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of LIV-GAMMA SN Inj.10% administered for 2 days in adult subjects with primary immune thrombocytopenia (ITP). The primary objective of this study is to determine the responder rate. A response is defined as a platelet count of ≥30×10^9/L and at least a 2-fold increase of the baseline, confirmed on at least 2 separate occasions at least 7 days apart without bleeding. The secondary objectives are to evaluate the further efficacy assessments including time to response and duration of response, and the safety of LIV-GAMMA SN Inj.10%.

ELIGIBILITY:
Inclusion Criteria:

* Completed informed consent process
* Male or female aged ≥19 years
* Diagnosis of chronic ITP (≥12 months since diagnosis)
* Mean screening platelet count of <30×10^9/L from 3 qualifying platelet counts performed within 14 days before the start of treatment, with no individual platelet count above 35×10^9/L
* No other factors inducing ITP
* If the patient is taking corticosteroid, attenuated androgen, cyclophosphamide, azathioprine or other drugs for ITP, the treatment regimen and dose should be stable at least 1 month prior to screening and should be lasted during this study
* Females of child-bearing potential with a negative urine pregnancy test and who agree with contraception during this study

Exclusion Criteria:

* Patients who have allergy or hypersensitivity to blood products, blood-derived products, intravenous immunoglobulin (IVIg) or immunoglobulin G (IgG)
* Patients who have immunoglobulin A (IgA) deficiency
* Patients who were immunized with live attenuated vaccines within 12 months from the first administration of LIV-GAMMA SN Inj.10%
* Patients who had received IVIg or blood/blood-derived products within 1 month from the first administration of LIV-GAMMA SN Inj.10%
* Patients who had received other investigational products within 1 month from the first administration of LIV-GAMMA SN Inj.10%
* Patients who had received Rituximab within 3 months from the first administration of LIV-GAMMA SN Inj.10%
* Patients who were taking anticoagulants or other agents related to platelet function (e.g., Aspirin, other NSAID) at the time of screening
* Patients who are pregnant and nursing
* Patients who are positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) at the time of screening
* Patients who have 3-fold higher levels of alanine transaminase (ALT), aspartate transaminase (AST) than the upper limit of normal at the time of screening
* Patients who suffered from severe renal impairment (eGFR<30 mL/min/1.73 m^2 at the time of screening)
* Patients who had history of deep vein thrombosis (DVT) or thrombotic complications against IVIg therapy
* Patients who had history of neurovascular or cardiovascular disorders (e.g., Blood hyperviscosity, transient ischemic attack (TIA), stroke, other thromboembolism, unstable angina)
* Patients who have an ongoing history of acute or chronic condition that affect to the participation of this study
* Patients who have an ongoing history of medical condition inducing secondary immune deficiency (e.g., Leukemia, lymphoma, multiple myeloma, HIV infection, chronic or cyclic neutropenia (absolute neutrophil count<500/mm^3)
* Patients who are suffering from hypertension (systolic blood pressure>160 mmHg or diastolic blood pressure>100 mmHg)
* Patients who have hemoglobin level≤10 g/dL at the time of screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Responder rate (CR or R) | 28 days
  The rate of subjects with complete response (CR) defined as cases with a platelet count ≥100×10^9/L, confirmed on at least 2 separate occasions at least 7 days apart with an absence of bleeding or response (R) defined as cases with a platelet count ≥30×10^9/L and at least a 2-fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart with an absence of bleeding

SECONDARY OUTCOMES:
The percentage of subjects with complete response (CR) | 28 days
  The percentage of subjects with complete response (CR) defined as cases with a platelet count ≥100×10^9/L, confirmed on at least 2 separate occasions at least 7 days apart with an absence of bleeding
The percentage of subjects with response (R) | 28 days
  The percentage of subjects with response (R) defined as cases with a platelet count ≥30×10^9/L and at least a 2-fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart with an absence of bleeding
Time to response | 28 days
  The time from the treatment initiation to the day when complete response (CR) or response (R) is achieved
Duration of response | 28 days
  The time from the achievement of complete response (CR) or response (R) to the day when loss of complete response (CR) or response (R) is achieved
Bleeding | 28 days
  Bleeding assessment with ITP-BAT bleeding grading system
Adverse events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jong Wook Lee, MD, Study Chair — The Catholic University of Korea
Locations (11):
- South Korea (11):
  - Dong-A University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul